CLINICAL TRIAL: NCT04750096
Title: Respiratory Failure in Esophagectomy. Results After Implantation of Enhanced Recovery After Surgery Protocol.
Brief Title: Esophagectomy Enhanced Recovery After Surgery Protocol
Acronym: ERASE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Raquel Ferrandis Comes (Other)
Responsible Party: Sponsor-Investigator, Raquel Ferrandis Comes, Doctor, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Other Study IDs: ERASE 001
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Esophagectomy
Keywords: Esophagectomy; enhanced recovery after surgery; acute lung injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Esophagectomy post enhanced recovery after surgery: Patients undergoing esophagectomy due to oesophageal cancer under Enhanced Recovery After Surgery protocol.

SUMMARY:
Despite the important advances in anaesthesia and the implementation of perioperative care, pulmonary complications in esophagectomy reach figures of between 20 and 35%, and these complications are also closely associated with the mortality rate. Factors that have been associated with the development of respiratory failure in the literature include among others the presence of previous respiratory pathology, history of smoking, malnutrition and rescue surgery.

With the aim of improving morbimortality in patients undergoing esophagectomy, a multidisciplinary protocol based on the best scientific evidence at the present time has been implemented, with actions covering both the preoperative and postoperative areas. Based on this point, a prospective study has been designed that allows us to compare the incidence of respiratory failure before and after the implementation of the protocol.

DETAILED DESCRIPTION:
Esophageal carcinoma is the sixth leading cause of cancer death worldwide and the main treatment still remains oesophagectomy, a technique associated with a high morbidity and mortality rate. Despite the important advances in anaesthesia and the implementation of perioperative care, pulmonary complications in these patients reach figures of between 20 and 35%, and these complications are also closely associated with the mortality rate. Factors that have been associated with the development of respiratory failure in the literature include among others the presence of previous respiratory pathology, history of smoking, malnutrition and rescue surgery.

With the aim of improving morbimortality in patients undergoing oesophagectomy, a multidisciplinary protocol based on the best scientific evidence at the present time has been implemented, with actions covering both the preoperative and postoperative areas. Based on this point, a prospective study has been designed that allows us to compare the incidence of respiratory failure before and after the implementation of the protocol.

The secondary objectives are to analyse the changes produced in terms of morbimortality after the implementation of the protocol and the repercussion of these changes on the length of stay in the Resuscitation Unit.

To carry out this project, data obtained in the first instance from patients operated before the implementation of the enhanced recovery after surgery protocol will be compared with data obtained prospectively after the implementation of the protocol.

The data will be collected from the computerised and digitalised medical records of the patients on Orion Clinic® and Interspace intelligence Critical Care and Anesthesia, Philips ®. Patients operated on between 19 October 2020 and 19 October 2021 will be included consecutively. Prior to the operation, patients must sign an informed consent form to authorize the monitoring of their data during the first 30 days after the operation. These data will include:

* Days of stay
* Development or not of respiratory failure on initial admission, as well as the ventilatory therapy used (non-invasive and invasive) and days of mechanical ventilation
* Fluid balance at 24 hours
* Adequate completion of the protocol on a post-operative basis. The items of the protocol completed during the postoperative period will be detailed, taking into account the following points:

  1. Use of epidural analgesia
  2. Adequate pain control
  3. Realisation of neutral or negative balances
  4. Introduction of enteral nutrition by jejunostomy
  5. Performance of respiratory physiotherapy
  6. Use of high-flow nasal glasses with a minimum flow of 40 litres.
  7. Start of sedation on the second post-operative day
  8. Antithrombotic prophylaxis
* The need or not for new drains and the reason for their installation will also be collected in order to evaluate the effectiveness of the transhiatal drains included in our protocol.

Data regarding re-entry will be collected on

* Reason for re-entry
* Evolutionary day after surgery when readmission took place (day 1 being counted as the day of esophagectomy)
* Days in the Critical Care Unit
* Development or not of respiratory insufficiency, and in positive cases, requirement of invasive or non-invasive mechanical ventilation and days of therapy with it.

Finally, the morbidity and mortality variables will be collected:

* Respiratory complications: pleural effusion, atelectasis, pneumothorax, pneumonia, adult respiratory distress syndrome (ARDS).
* The development of complications other than respiratory ones.
* The need for reintervention and the underlying cause.
* If exits occur, as well as the cause of death in hospital or in the first 30 days after surgery.

The data will be analysed using Statistical Package for the Social Sciences software ® (version 12).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone esophagectomy due to neoplastic causes
* Ages between 18 and 90
* Programmed surgery

Exclusion Criteria:

* Caustic esophagitis
* Esophagectomy for stomach cancer
* Congenital oesophageal malformations

  * Respiratory failure at the time of surgery
  * Re-interventions of esophagectomy
* Unexpected intraoperative surgical problems

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing esophagectomy due to oesophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative respiratory failure | 1 month
  Post-operative respiratory failure in esophagectomy after introduction of Enhanced Recovery After Surgery protocol

SECONDARY OUTCOMES:
Other morbidity | 1 month
  Analyse changes in terms of morbidity and mortality different from respiratory failure following the implementation of the protocol. It will allow us to know the impact of the measures carried out on complications and mortality.
Stay at ICU | 1 month
  Changes produced in the resuscitation stay after the Enhanced Recovery After Surgery protocol.
Main predisposing factors | 1 month
  Main predisposing factors for the development of respiratory insufficiency.
Respiratory failure as a prognostic factor | 1 month
  Analyse the presence of respiratory failure as a prognostic factor. This allows us to know the impact of respiratory failure on the evolution of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- La Fe University and Polytechnic Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Low DE, Kuppusamy MK, Alderson D, Cecconello I, Chang AC, Darling G, Davies A, D'Journo XB, Gisbertz SS, Griffin SM, Hardwick R, Hoelscher A, Hofstetter W, Jobe B, Kitagawa Y, Law S, Mariette C, Maynard N, Morse CR, Nafteux P, Pera M, Pramesh CS, Puig S, Reynolds JV, Schroeder W, Smithers M, Wijnhoven BPL. Benchmarking Complications Associated with Esophagectomy. Ann Surg. 2019 Feb;269(2):291-298. doi: 10.1097/SLA.0000000000002611. PMID 29206677
- [Background] Takeuchi H, Miyata H, Ozawa S, Udagawa H, Osugi H, Matsubara H, Konno H, Seto Y, Kitagawa Y. Comparison of Short-Term Outcomes Between Open and Minimally Invasive Esophagectomy for Esophageal Cancer Using a Nationwide Database in Japan. Ann Surg Oncol. 2017 Jul;24(7):1821-1827. doi: 10.1245/s10434-017-5808-4. Epub 2017 Feb 21. PMID 28224366
- [Background] van Adrichem EJ, Meulenbroek RL, Plukker JT, Groen H, van Weert E. Comparison of two preoperative inspiratory muscle training programs to prevent pulmonary complications in patients undergoing esophagectomy: a randomized controlled pilot study. Ann Surg Oncol. 2014 Jul;21(7):2353-60. doi: 10.1245/s10434-014-3612-y. Epub 2014 Mar 7. PMID 24604584
- [Background] Armestar F, Mesalles E, Font A, Arellano A, Roca J, Klamburg J, Fernandez-Llamazares J. [Serious postoperative complications after esophagectomy for esophageal carcinoma: analysis of risk factors]. Med Intensiva. 2009 Jun-Jul;33(5):224-32. doi: 10.1016/s0210-5691(09)71756-5. Spanish. PMID 19624996
- [Background] Liu F, Wang W, Wang C, Peng X. Enhanced recovery after surgery (ERAS) programs for esophagectomy protocol for a systematic review and meta-analysis. Medicine (Baltimore). 2018 Feb;97(8):e0016. doi: 10.1097/MD.0000000000010016. PMID 29465538
- [Background] Findlay JM, Gillies RS, Millo J, Sgromo B, Marshall RE, Maynard ND. Enhanced recovery for esophagectomy: a systematic review and evidence-based guidelines. Ann Surg. 2014 Mar;259(3):413-31. doi: 10.1097/SLA.0000000000000349. PMID 24253135
- [Background] Lagarde SM, Maris AK, de Castro SM, Busch OR, Obertop H, van Lanschot JJ. Evaluation of O-POSSUM in predicting in-hospital mortality after resection for oesophageal cancer. Br J Surg. 2007 Dec;94(12):1521-6. doi: 10.1002/bjs.5850. PMID 17929231
- [Background] van der Sluis PC, Schizas D, Liakakos T, van Hillegersberg R. Minimally Invasive Esophagectomy. Dig Surg. 2020;37(2):93-100. doi: 10.1159/000497456. Epub 2019 May 16. PMID 31096214
- [Background] Lv L, Hu W, Ren Y, Wei X. Minimally invasive esophagectomy versus open esophagectomy for esophageal cancer: a meta-analysis. Onco Targets Ther. 2016 Oct 31;9:6751-6762. doi: 10.2147/OTT.S112105. eCollection 2016. PMID 27826201
- [Background] Palanivelu C, Prakash A, Senthilkumar R, Senthilnathan P, Parthasarathi R, Rajan PS, Venkatachlam S. Minimally invasive esophagectomy: thoracoscopic mobilization of the esophagus and mediastinal lymphadenectomy in prone position--experience of 130 patients. J Am Coll Surg. 2006 Jul;203(1):7-16. doi: 10.1016/j.jamcollsurg.2006.03.016. PMID 16798482
- [Background] Kinugasa S, Tachibana M, Yoshimura H, Ueda S, Fujii T, Dhar DK, Nakamoto T, Nagasue N. Postoperative pulmonary complications are associated with worse short- and long-term outcomes after extended esophagectomy. J Surg Oncol. 2004 Nov 1;88(2):71-7. doi: 10.1002/jso.20137. PMID 15499604
- [Background] Ferguson MK, Celauro AD, Prachand V. Prediction of major pulmonary complications after esophagectomy. Ann Thorac Surg. 2011 May;91(5):1494-1500; discussion 1500-1. doi: 10.1016/j.athoracsur.2010.12.036. PMID 21524462
- [Background] Kobayashi S, Kanetaka K, Nagata Y, Nakayama M, Matsumoto R, Takatsuki M, Eguchi S. Predictive factors for major postoperative complications related to gastric conduit reconstruction in thoracoscopic esophagectomy for esophageal cancer: a case control study. BMC Surg. 2018 Mar 6;18(1):15. doi: 10.1186/s12893-018-0348-9. PMID 29510754
- [Background] Biere SS, van Berge Henegouwen MI, Bonavina L, Rosman C, Roig Garcia J, Gisbertz SS, van der Peet DL, Cuesta MA. Predictive factors for post-operative respiratory infections after esophagectomy for esophageal cancer: outcome of randomized trial. J Thorac Dis. 2017 Jul;9(Suppl 8):S861-S867. doi: 10.21037/jtd.2017.06.61. PMID 28815084
- [Background] Law S, Wong KH, Kwok KF, Chu KM, Wong J. Predictive factors for postoperative pulmonary complications and mortality after esophagectomy for cancer. Ann Surg. 2004 Nov;240(5):791-800. doi: 10.1097/01.sla.0000143123.24556.1c. PMID 15492560
- [Background] Ferguson MK, Durkin AE. Preoperative prediction of the risk of pulmonary complications after esophagectomy for cancer. J Thorac Cardiovasc Surg. 2002 Apr;123(4):661-9. doi: 10.1067/mtc.2002.120350. PMID 11986593
- [Background] Choi H, Cho JH, Kim HK, Choi YS, Kim J, Zo JI, Shim YM, Jeon K. Prevalence and clinical course of postoperative acute lung injury after esophagectomy for esophageal cancer. J Thorac Dis. 2019 Jan;11(1):200-205. doi: 10.21037/jtd.2018.12.102. PMID 30863589
- [Background] Shirinzadeh A, Talebi Y. Pulmonary Complications due to Esophagectomy. J Cardiovasc Thorac Res. 2011;3(3):93-6. doi: 10.5681/jcvtr.2011.020. Epub 2011 Aug 20. PMID 24250962